CLINICAL TRIAL: NCT02589717
Title: An Open-Label, Multicenter, Expanded Access Program for Atezolizumab in Patients With Locally Advanced or Metastatic Urothelial Carcinoma After Failure With Platinum-Containing Chemotherapy.
Brief Title: An Expanded Access Study of Atezolizumab in Participants With Locally Advanced or Metastatic Urothelial Carcinoma After Failure With Platinum-Containing Chemotherapy
Status: Approved for marketing | Type: Expanded Access
Sponsor: Genentech, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: ML29725
Record Dates: First submitted 2015-10-16; First posted 2015-10-28 (Estimated); Last update posted 2016-11-02 (Estimated); Status verified 2016-11

CONDITIONS: Urothelial Carcinoma
MeSH Terms: conditions — Carcinoma, Transitional Cell | interventions — atezolizumab

INTERVENTIONS:
Drug: Atezolizumab [TECENTRIQ] — Atezolizumab 1200 mg will be administered by IV infusion q3w. Initial IV infusion will be given over 60 minutes and subsequent infusions will be given over 30 minutes.

SUMMARY:
This is an open-label, multicenter, single-arm, expanded access program (EAP) designed to provide atezolizumab access to participants with locally advanced or metastatic urothelial carcinoma that has progressed on, or is intolerant to, a platinum-containing chemotherapy regimen.

ELIGIBILITY:
Inclusion Criteria:

* Able to comply with the study protocol, in the investigator's judgment
* Histologically or cytologically documented locally advanced or metastatic urothelial carcinoma (including renal pelvis, ureters, urinary bladder, and urethra)
* Disease progression during or following treatment with at least one platinum-containing regimen (e.g., gemcitabine and cisplatin [GC], methotrexate, vinblastine, doxorubicin, and cisplatin [MVAC], carboplatin and gemcitabine [CarboGem], etc.) for inoperable locally advanced or metastatic urothelial carcinoma or disease recurrence
* Eastern Cooperative Oncology Group (ECOG) Performance Status of 0, 1, or 2
* Life expectancy >/= 12 weeks
* Adequate hematologic and end-organ function, defined by laboratory results obtained within 14 days prior to the first study treatment
* For women who are not postmenopausal (>/= 12 months of non-therapy-induced amenorrhea) or surgically sterile (absence of ovaries and/or uterus): agreement to remain abstinent or use single or combined non-hormonal contraceptive methods that result in a failure rate of <1% per year during the treatment period and for at least 90 days after the last dose of study drug

Exclusion Criteria:

* Treatment with any other investigational agent or participation in another clinical trial with therapeutic intent within 28 days prior to enrollment
* Treatment with chemotherapy 14 days prior to enrollment; however, participants may be re-screened after the 14-day washout period
* Treatment with radiotherapy 7 days prior to enrollment; however, participants may be re-screened after the 14-day washout period
* Known primary central nervous system (CNS) malignancy or symptomatic CNS metastases
* Pregnant or lactating, or intending to become pregnant during the study
* Significant cardiovascular disease, such as New York Heart Association cardiac disease (Class II or greater), myocardial infarction within 3 months prior to randomization, unstable arrhythmias, or unstable angina
* Severe infections within 4 weeks prior to enrollment, including, but not limited to, hospitalization for complications of infection, bacteremia, or severe pneumonia
* Received therapeutic oral or intravenous (IV) antibiotics within 14 days prior to enrollment; however, participants may be re-screened after the 14-day washout period
* Major surgical procedure within 4 weeks prior to enrollment or anticipation of need for a major surgical procedure during the course of the study other than for diagnosis
* History of severe allergic, anaphylactic, or other hypersensitivity reactions to chimeric or humanized antibodies or fusion proteins
* Known hypersensitivity or allergy to biopharmaceuticals produced in Chinese hamster ovary cells or any component of the atezolizumab formulation
* Any other diseases, metabolic dysfunction, physical examination finding, or clinical laboratory finding giving reasonable suspicion of disease or a condition that contraindicates the use of the investigational drug or renders the participant at high risk for treatment complications
* Participants with active hepatitis B
* Active tuberculosis
* Administration of a live, attenuated vaccine within 4 weeks prior to enrollment or anticipation that such a live, attenuated vaccine will be required during the study
* Treatment with systemic immunostimulatory agents (including, but not limited to, interferons or IL-2) within 4 weeks or five half-lives of the drug, whichever is shorter, prior to enrollment
* Treatment with systemic corticosteroids or other systemic immunosuppressive medications (including, but not limited to, prednisone, dexamethasone, cyclophosphamide, azathioprine, methotrexate, thalidomide, and anti-tumor necrosis factor [anti-TNF] agents) within 2 weeks prior to enrollment or anticipated requirement for systemic immunosuppressive medications during the trial

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 2015-11; Primary Completion 2016-08 (Actual); Study Completion 2016-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Genentech, Inc.
Locations (38):
- United States (38):
  - Scottsdale, Arizona
  - Tucson, Arizona
  - Duarte, California
  - Oakland, California
  - Stanford, California
  - Denver, Colorado
  - New Haven, Connecticut
  - West Hartford, Connecticut
  - Miami Beach, Florida
  - Tampa, Florida
  - Harvey, Illinois
  - Springfield, Illinois
  - Goshen, Indiana
  - Indianapolis, Indiana
  - Sioux City, Iowa
  - Louisville, Kentucky
  - New Orleans, Louisiana
  - Boston, Massachusetts
  - Ann Arbor, Michigan
  - Detroit, Michigan
  - Saint Cloud, Minnesota
  - Jackson, Mississippi
  - St Louis, Missouri
  - Albuquerque, New Mexico
  - Abany, New York
  - New York, New York
  - Rochester, New York
  - Columbus, Ohio
  - Eugene, Oregon
  - Easton, Pennsylvania
  - Philadelphia, Pennsylvania
  - Pittsburgh, Pennsylvania
  - Charleston, South Carolina
  - Houston, Texas
  - San Antonio, Texas
  - Charlottesville, Virginia
  - Norfolk, Virginia
  - Spokane, Washington